CLINICAL TRIAL: NCT06796933
Title: Effect of Bioptron on Scar Formation After Cesarean Section: a Randomized Controlled Trial
Brief Title: Effect of Bioptron on Scar Formation After Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghadeer Abdelazzim Mostafa, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005315
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cesarean Section

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silicone-based products group (Active Comparator): The participants will be treated with cosmetic creams such as Silicone-based products, (silicone gels for 1 month).
  Interventions: Other: Silicon based products (silicon gel)
- Bioptron and Silicone-based products group (Experimental): The participants will be treated by polarized light therapy (Bioptron) for 15 minutes, 3 sessions per week, in addition to the cosmetic creams (Silicone-based products; silicone gels) for one month.
  Interventions: Other: Silicon based products (silicon gel); Device: Bioptron (polarized light therapy)

INTERVENTIONS:
Other: Silicon based products (silicon gel) — The participants will be treated with cosmetic creams such as Silicone-based products (silicone gels twice a day) for one month.
Device: Bioptron (polarized light therapy) — The participants will be treated by polarized light therapy (Bioptron) for 15 minutes, 3 sessions per week, for one month.
  Arms: Bioptron and Silicone-based products group

SUMMARY:
The purpose of the study will be to determine the effect of polarized light therapy (Bioptron) on scar formation after a cesarean section.

DETAILED DESCRIPTION:
Cesarean deliveries are among the most frequently performed surgical procedures for women worldwide, with their prevalence increasing globally, especially in developing nations like Egypt.

A scar is a natural outcome of the healing process following a wound. Complaints associated with scars can lead to both physical discomfort and psychological challenges. Enhanced healing of CS scars could lead to better postoperative outcomes, reducing complications such as infection, pain, and restricted mobility. These aspects of recovery are often neglected, as noted by.

This study will be the first to specifically examine the effects of Bioptron light therapy on CS scar formation. While previous research has shown the benefits of this therapy on scars from various operations, none have focused on CS scars. By investigating this innovative, non-invasive treatment approach, the study aims to fill a critical gap in existing research and offer valuable insights into managing and improving postoperative recovery for CS patients.

ELIGIBILITY:
Inclusion Criteria:

* The participants' ages will be ranged from 20-30 years old.
* Their body mass index (BMI) will not exceed 30 kg/m2.
* They will be primipara and having abdominal scar after CS.
* The scar age will be extended from 6 weeks to 6 months.
* All women will be medically stable when attending the study.

Exclusion Criteria:

* Pregnant women or women planning to become pregnant during the study period.
* Women having diabetes mellitus.
* Women taking immunosuppressant drugs.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-01-27 (Estimated); Primary Completion 2025-03-18 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The Patient and Observer Scar Assessment Scale (POSAS) | 4 weeks
  It is a comprehensive tool designed to evaluate scar quality from both the patient's and the observer's perspectives before and after treatment for all participants in both groups. This scale includes two separate assessments: one completed by the patient and the other by the healthcare professional observing the scar. Each part of the scale assesses different aspects of the scar, providing a holistic view of its impact and severity.
  Each scale assesses six scar characteristics: the observer evaluates vascularization, pigmentation, thickness, surface roughness, pliability, and surface area, while the patient rates pain, pruritus, color, thickness, relief, and pliability. All items are scored on a 10-point scale, with 1 indicating 'normal skin' and 10 representing the 'worst imaginable scar.' Higher total scores indicate poorer scar quality
Vancouver scar scale | 4 weeks
  The Vancouver Scar Scale (VSS) is a widely used tool for assessing the quality and severity of scars before and after treatment for all participants in both groups. The VSS helps clinicians objectively measure the effectiveness of treatments and track changes in scar characteristics over time The VSS rated the scars according to four parameters: vascularity, pigmentation, pliability, and height. Each parameter contained ranked subscales that may be summed to obtain a total score ranging from 0 (representing normal skin) to 13 (representing the worst scar imaginable).

SECONDARY OUTCOMES:
Adheremeter | 4 weeks
  The modified adheremeter is a plastic sheet with a radius of 4.6 cm, and concentric circles 2 mm apart. It is described as a measurement tool for assessing the extensibility of peripheral surgical scars; it is utilized in evaluating the extensibility of abdominal tissue. Skin mobility at specific points is measured in four directions, and the area of mobility is then calculated. It was reported to have excellent intra-rater reliability when using this method on abdominal tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Assar, Professor, Study Director — Benha University; Mohamed Awad, Professor, Study Chair — Cairo University
Locations (1):
- Ghadeer Abdelazim Mostafa, Banhā, Egypt